CLINICAL TRIAL: NCT02979327
Title: Cardiovascular Effects of Adderall in Healthy Adults. A Randomized Clinical Trial.
Brief Title: Cardiovascular Effects of Adderall in Healthy Adults.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Anna Svatikova, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 16-004743
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Hemodynamics; Cardiovascular System
MeSH Terms: interventions — Adderall

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adderall first, then Placebo (Experimental): Participants will receive an Adderall capsule at the first study visit, then a Placebo capsule at the second study visit.
  Interventions: Drug: Adderall capsule; Drug: Placebo capsule
- Placebo first, then Adderall (Experimental): Participants will receive a Placebo capsule at the first study visit, then an Adderall capsule at the second study visit.
  Interventions: Drug: Adderall capsule; Drug: Placebo capsule

INTERVENTIONS:
Drug: Adderall capsule — 25 mg orally one time
Drug: Placebo capsule — Looks exactly like the study drug, but it contains no active ingredient. Taken one time.

SUMMARY:
This study is designed to investigate the cardiovascular response (blood pressure, heart rate, electrocardiographic response and blood vessel reactivity response) to taking Adderall in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age and older
2. Healthy subjects without known cardiovascular disease, thyroid disease or documented mental health illness
3. Subjects who are on no medications
4. Subjects with no prior history of regular amphetamine use, and non-prescription stimulants
5. Nonsmokers

Exclusion Criteria

1. Subjects with known cardiovascular disease, thyroid disease
2. Subjects with history of psychotic disorders/mental health illness, including but not limited to anxiety, depression, bipolar disorder; history of substance abuse or dependence
3. Subjects currently taking medications
4. Prior history of regular amphetamine use, or non-prescription stimulants
5. Smokers
6. Pregnant subjects
7. Known lactose intolerance (due to presence of lactose in the prepared medication)
8. Family history of sudden cardiac death

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Svatikova, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adderall First, Then Placebo: Subjects received an Adderall capsule at the first study visit, then they received a Placebo capsule at the second study visit.
  Adderall capsule: 25 mg orally one time
  Placebo capsule: Looks exactly like the study drug, but it contains no active ingredient. Taken one time.
- Placebo First, Then Adderall: Subjects received a Placebo capsule at the first study visit, then they received an Adderall capsule at the second study visit.
  Adderall capsule: 25 mg orally one time
  Placebo capsule: Looks exactly like the study drug, but it contains no active ingredient. Taken one time.
Period: First Intervention
Arm/Group | Adderall First, Then Placebo | Placebo First, Then Adderall
Started | 17 | 13
Completed | 16 | 13
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Second Intervention
Arm/Group | Adderall First, Then Placebo | Placebo First, Then Adderall
Started | 16 | 13
Completed | 16 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adderall First, Then Placebo | Placebo First, Then Adderall | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (5) | 28 (6) | 27 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 6 | 8 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure (top number of blood pressure reading)
Time Frame: Baseline and 3 hours
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Adderall: Subjects who received an Adderall capsule at either the first or second study visit
  Adderall capsule: 25 mg orally one time
- Placebo: Subjects who received a Placebo capsule at either the first or second study visit
  Placebo capsule: Looks exactly like the study drug, but it contains no active ingredient. Taken one time.
Arm/Group | Adderall | Placebo
Number analyzed (Participants) | 29 | 29
mmHg
  baseline | 116 (2) | 116 (2)
  3 hours | 126 (2) | 115 (2)

2. Primary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure (bottom number of blood pressure reading)
Time Frame: Baseline and 3 hours
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Adderall | Placebo
Number analyzed (Participants) | 29 | 29
mmHg
  baseline | 72 (2) | 72 (1)
  3 hours | 78 (2) | 71 (2)

3. Primary Outcome: Mean Arterial Pressure (MAP)
Description: Mean arterial pressure (MAP) is a measure of the average blood pressure in the large arteries. It accounts for the blood flow and resistance. Measured in millimeters of mercury (mmHg)
Time Frame: Baseline and 3 hours
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Adderall | Placebo
Number analyzed (Participants) | 29 | 29
mmHg
  baseline | 87 (2) | 86 (1)
  3 hours | 94 (2) | 86 (2)

4. Primary Outcome: Heart Rate
Description: Number of beats per minute
Time Frame: Baseline and 3 hours
Measure: Mean (Standard Error); unit: beats/min
Arm/Group | Adderall | Placebo
Number analyzed (Participants) | 29 | 29
beats/min
  baseline | 60 (2) | 59 (2)
  3 hours | 70 (3) | 61 (2)

5. Secondary Outcome: Plasma Norepinephrine
Description: Measurement of norepinephrine levels in the plasma. The normal range is 70 to 1700 pg/mL
Time Frame: baseline and 3 hours
Population: Data was not collected nor analyzed for four subjects in each arm
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Adderall | Placebo
Number analyzed (Participants) | 25 | 25
pg/ml
  baseline | 215 (15) | 217 (23)
  3 hours | 301 (14) | 227 (17)

ADVERSE EVENTS:
Time Frame: Adverse events were collected on all subjects from baseline to end of study, approximately 2 months.
Arm/Group | Adderall | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 1/29 | 2/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adderall (N=29) | Placebo (N=29)
Lightheadedness (General disorders) | 0 | 1
Headache (General disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Tingling in fingers, toes, face (Nervous system disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT02979327/Prot_SAP_000.pdf